CLINICAL TRIAL: NCT03516955
Title: Observational Study of Superstat® (Rosuvastatin) in Hypercholesterolemia Patients in Lebanon
Brief Title: Efficacy and Safety of a Generic Rosuvastatin in a Real-world Setting
Status: Completed | Type: Observational
Sponsor: Hikma Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: SPS-LBN-2014-05
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Primary Hypercholesterolemia
Keywords: Superstat; Rosuvastatin; Statins; LDL-C; Cholesterol; Hypercholesterolemia; Dyslipidemia; Coronary Artery Disease; Cardiovascular Disease
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias; Coronary Artery Disease; Cardiovascular Diseases | interventions — Rosuvastatin Calcium; superstat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rosuvastatin — Superstat ® Tablets 10mg, 20mg
  Other Names: Superstat ®

SUMMARY:
This study assessed the safety and efficacy of generic Rosuvastatin in reducing plasma low density lipoprotein (LDL) cholesterol in Lebanese adult patients (18 years or older) with dyslipidemia for both primary and secondary prevention based on their total cardiovascular risk. No visits or interventions, additional to the routine clinical practice, were requested or performed.

DETAILED DESCRIPTION:
An observational, multicenter, prospective study of Lebanese adult (18 years or older) hypercholesterolemic patients administered generic Rosuvastatin (Superstat®).

Eligible newly diagnosed hypercholesterolemic patients took generic Rosuvastatin as prescribed by their treating physician. Assigning patients to generic Rosuvastatin was decided within the current practice and medical indication and was independent from the recruitment into the study.

Patients were followed-up at the clinic as per the standard practice of care. Each patient was followed-up for a period of 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Patients with dyslipidemia requiring statin therapy according to CV risk factors as per the ESC/EAS 2011 guidelines for primary or secondary prevention
* Patients provided written informed consent

Exclusion Criteria:

* Age <18 years
* Statin use in the past 3 months
* Any contraindication to HMG-CoA reductase inhibitors
* Co-administration of non-statin lipid lowering agent (ezitimibe, fibrates, niacin, omega 3)
* Conditions which may cause secondary dyslipidemia
* Any of the following abnormal laboratory tests:

TG level of > 400 mg/dL, Abnormal liver enzymes (AST or ALT) ≥ 3 ULN, Abnormal serum creatine kinase (CK) > 5 ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from 24 cardiology, endocrinology and general practitioner outpatient clinics in Lebanon
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Percent change in mean low-density lipoproteins (LDL-C) | 2 months

SECONDARY OUTCOMES:
Percent change in mean total cholesterol, triglycerides, high density lipoprotein (HDL-C) | 2 months
Proportion of patients who meet their target (LDL-C) | 2 months
Incidence rate of adverse events (AEs) in association with generic rosuvastatin | 2 months
  Rate of AEs which might include the worsening in baseline medical conditions, the occurrence of new conditions, or a significant change in vital signs or laboratory values.